CLINICAL TRIAL: NCT02462031
Title: A Randomized, Double-blind, Placebo-controlled, Single or Multiple Ascending Dose Phase I Clinical Trial to Evaluate the Safety, Tolerability, PK, PK-PD Relation of KD101 in the Fed State in Obese or Overweight Subjects
Brief Title: To Evaluate the Safety, Tolerability, PK, PK-PD Relation of KD101 in the Fed State in Obese or Overweight Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kwang Dong Pharmaceutical co., ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: KD101-102
Record Dates: First submitted 2015-05-06; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KD101 (Experimental)
  Interventions: Drug: KD101
- KD101 placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: KD101 — 200mg, 400mg, 800mg, 1400mg
  Other Names: KD101 soft capsule 200mg
  Arms: KD101
Drug: placebo — 200mg, 400mg, 800mg
  Other Names: KD101 soft capsule 200mg placebo
  Arms: KD101 placebo

SUMMARY:
To Evaluate the safety, tolerability and pharmacokinetic property after KD101 multiple oral dosing in the fed state in obese or overweight subjects.

DETAILED DESCRIPTION:
dose block-randomized, double-blinded, placebo controlled, single or multiple ascending dose study. AEs, PE, Vital signs, ECGs and Clinical lab tests

* Part I : multiple dose study (KD101 or placebo) / male and female
* Part II : single dose study (KD101) / male only

ELIGIBILITY:
Inclusion Criteria:

* Male or Female adults aged 20 to 55 at screening (Part II : Male adults aged 20 to 55 at screening)
* Healthy volunteer whose BMI ≥ 27 (Part II : Healthy volunteer whose BMI ≥ 18)
* Female who are not pregnancy possibility or Male/Female who can abstinence or contraception during clinical trials

Exclusion Criteria:

* Subjects who had clinically significant disease history (liver,kidney,nervous,pulmonary,endocrinal,urinary,cardiovascular,musculoskeletal,mental system,blood,tumor) or diagnosed within 1 month from screening
* Subjects who had gastrointestinal disease(Crohn's disease, ulcer, acute/chronic pancreatitis) that affect the absorption of test drug or gastrointestinal operation (However, appendectomy, herniotomy induced by acute appendicitis are excluded)
* Subjects who had following history. [myocardial infarction (diagnosed by cardiac enzyme and/or diagnostic ECG), cerebral infarction/stroke, arrhythmia needed to medical treatment, unstable angina, pulmonary hypertension]
* Subjects who had positive result to Human Immunodeficiency Virus, Hepatitis B virus, Hepatitis C virus during screening
* Subjects who had allergy history (ex. allergy for aspirin, antibiotics, etc) or had clinically-significant allergy
* Subjects whose systolic BP was <85mmHg or >145mmHg, or diastolic BP was <50mmHg or >95mmHg, or pulse was >100/min after 3 minute-seating position. (BP can be re-measured twice at leat 5 minute-interval)
* Subjects who would take prescribed/oriental drug(within 2 weeks from the first dosing day) or OTC drug or vitamines (within 1 weeks from the first dosing day)
* Subjects who drink over than 21 unit (1 unit = 10g of pure alcohol) or cannot quit drinking alcohol during clinical trial period
* Subjects who ate following food within 2 days from the first dosing day or cannot quit following food [grapefruit-contain food, caffein-contain food(coffee, green tea, black tea, soft drink, coffee milk, energy drink)]
* Subjects who didn't agree contraception
* Subjects who didn't agree to quit smoke
* Subjects who donated his/her blood within 2 months (whole blood) / 1 month (apheresis) or who took transfusion within 1 month
* Subjects who participated another clinical trials within 3 months from first dosing day. (The clinical trial completion day is defined as the last dosing day of past clinical trial)
* Subjects who are not adequate to this trial by lab examination and another reasons
* Subjects who weighed loss more than 5kg in 3 months

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters - Cmax | up to 4 weeks
  Cmax (Maximum concentration of drug in plasma)

SECONDARY OUTCOMES:
Pharmacodynamic parameters - PBMCs | up to 4 weeks
  PBMC (Peripheral blood mononuclear cell)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Lee, Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea